CLINICAL TRIAL: NCT05969028
Title: First Responder Airway & Compression Rate Trial (FACT Study)
Brief Title: First Responder Airway & Compression Rate Trial
Acronym: FACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Thomas Rea, Professor, School of Medicine, University of Washington
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00014110
Record Dates: First submitted 2023-05-19; First posted 2023-08-01 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: Airway Management; CPR; Emergency Medical Services; Basic Life Support
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest | interventions — Airway Management; Cardiopulmonary Resuscitation

STUDY DESIGN:
Intervention Model Description: We propose a factorial-design, cluster randomized controlled trial. In brief, this means that two interventions (the type of rescue breathing treatment and chest compression rate) will be studied in the same patient; and that randomizing patients to these treatments will switch over various time periods between groups of fire departments in King County. That is, some fire departments will be performing BVM with a compression rate of 100 compressions per minute over a specified time period, and will thereafter switch to the i-gel and a different chest compression rate for a specified time period.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Airway Strategy (Active Comparator): Each of 28 first responder EMS agencies in King County will be randomly assigned to treat with either the BVM or i-gel for airway strategy
  Interventions: Device: igel
- Compression Rate (Active Comparator): Each of 28 first responder EMS agencies in King County will be randomly assigned with one of the three chest compression rates (100 vs 110 vs 120) at the outset.
  Interventions: Procedure: Compression Rate

INTERVENTIONS:
Device: igel — First responder ventilation strategy. First responders in King County routinely use the BVM as part of core treatment of SCA. As part of EMS training, we have introduced a training module for use of the igel in simulated resuscitation, which has been enthusiastically accepted by EMS leadership and providers. The i-gel is already successfully practiced by BLS providers in a number of other communities and challenges in training and clinical application will be monitored, but not anticipated.
  Other Names: airway management; Bag Valve Mask
  Arms: Airway Strategy
Procedure: Compression Rate — Compression rates. The EMS system routinely measures EMS CPR performance and specifically the chest compression rate using information derived and electronically recorded from defibrillator patches. As detailed in the Background section, this CPR surveillance activity highlights the variability of compression rates across the guideline-directed range of 100-120 compressions per minute. In addition our CPR surveillance indicates that a metronome can be used to obtain and maintain a specific compression rate within the parameters specified by this trial. This will be the tool used to guide compliance with the assigned chest compression rate by on-scene providers.
  Other Names: CPR
  Arms: Compression Rate

SUMMARY:
The First responder Airway & Compression rate Trial (FACT) Study will address basic life support (BLS) treatments administered by Emergency Medical Services (EMS) first responders to patients who suffer a sudden circulatory (pulseless) collapse, referred to as sudden out-of-hospital cardiac arrest (SCA). The investigators propose a randomized controlled trial among persons who suffer SCA to compare these two rescue breathing approaches (standard Bag Valve Mask vs i-gel) along with evaluating a more precise chest compression rate within the range of 100-120 compressions per minute during CPR. Importantly, each of these treatments fall within established resuscitation guidelines and are already administered as part of standard care in clinical practice. Thus this proposed trial will essentially be comparing one standard-of-care treatment against another standard-of-care treatment.

The study will address two primary aims:

Aim 1: To compare survival to hospital discharge between SCA patients randomized to BVM versus the i-gel for rescue breathing. The hypothesis is that treatment with i-gel will result in a higher rate of survival to hospital discharge than BVM.

Aim 2: To compare survival to hospital discharge between SCA patients randomized to chest compression rates of 100 versus 110 versus 120 per minute. The hypothesis is that treatment with 100 chest compressions per minute will result in a higher rate of survival to hospital discharge than compression rates of 110 or 120 per minute.

DETAILED DESCRIPTION:
The First responder Airway & Compression rate Trial (FACT) Study will address basic life support (BLS) treatments administered by EMS first responders to patients who suffer a sudden circulatory (pulseless) collapse, referred to as sudden out-of-hospital cardiac arrest (SCA). The current standard of practice for first responder CPR includes chest compressions at a rate of 100-120 compressions per minute combined with rescue breathing using either a bag valve mask (BVM) or a type of oral airway called an i-gel. During rescue breathing with a BVM, a mask is attached to a breathing bag and placed over the patient's face. The BVM provides oxygen and clears carbon dioxide out of the lungs by blowing air through the patient's mouth. Alternatively, the i-gel consists of a short tube which is inserted in the back of the patient's throat. This tube blows oxygen more directly into the lungs, bypassing the mouth itself. Each of these breathing methods is considered standard of care treatment by EMS first responders. Standard of care means each method is commonly used to treat patients in cardiac arrest and is performed regularly, depending upon the community in which the cardiac arrest has occurred. The other component of CPR is chest compressions. The American Heart Association has recommended a chest compression rate during CPR of between 100-120 compressions per minute, but has not specified an ideal exact compression rate within this range. Scientific studies in both animals and clinical studies have shown that these different standard-of-care approaches to ventilation and the compression rate can produce different physiologic effects (such as the adequacy of rescue breathing and blood flow) that could impact clinical outcome. The investigators propose a randomized controlled trial among persons who suffer SCA to compare these two rescue breathing approaches along with evaluating a more precise chest compression rate within the range of 100-120 compressions per minute during CPR. Importantly, each of these treatments fall within established resuscitation guidelines and are already administered as part of standard care in clinical practice. Thus this proposed trial will essentially be comparing one standard-of-care treatment against another standard-of-care treatment.

The study will address two primary aims:

Aim 1: To compare survival to hospital discharge between SCA patients randomized to BVM versus the i-gel for rescue breathing. The hypothesis is that treatment with i-gel will result in a higher rate of survival to hospital discharge than BVM.

Aim 2: To compare survival to hospital discharge between SCA patients randomized to chest compression rates of 100 versus 110 versus 120 per minute. The hypothesis is that treatment with 100 chest compressions per minute will result in a higher rate of survival to hospital discharge than compression rates of 110 or 120 per minute.

ELIGIBILITY:
Inclusion Criteria:

* Adults suffering out-of-hospital non-traumatic SCA in Seattle and greater King County in whom resuscitation will be attempted by first responding EMS personnel.

Exclusion Criteria:

* if advanced paramedic providers are first on-scene and have already initiated advanced life support (ALS) procedures,
* a written advance directive (do not attempt resuscitation orders),
* traumatic arrest (blunt, penetrating, burn),
* known prisoner,
* known pregnancy,
* other protected populations (pediatrics),
* pre-existing tracheostomy,
* recipients of mechanical ventilator support, or
* presence of an "opt out" bracelet to not be enrolled in clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4200 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Survival to Hospital Discharge | This outcome typically occurs days to weeks after Cardiac Arrest Event. The study will monitor for this outcome for 6 months following the cardiac arrest event.
  The outcome will compare the proportion of subjects who survive to be discharged from the hospital. The outcome is an endorsed outcome by the Utstein guidelines and a common primary outcome in clinical resuscitation studies.

SECONDARY OUTCOMES:
Return to Spontaneous Circulation (ROSC) | This outcome occurs within minutes of the cardiac arrest event. The outcome will be monitored for 1 day from the time of cardiac arrest.
  This outcome provides a proximal outcome of the potential differential effectiveness of the study interventions.
Survival with favorable neurological function (CPC 1-2) | This outcome typically occurs days to weeks after Cardiac Arrest Event. The study will monitor for this outcome for 6 months following the cardiac arrest event.
  This outcome will compare the proportion of subjects who survive to be discharged from the hospital who have favorable functional status as determined by the Cerebral Performance Category. This outcome is an endorsed outcome measure by the Utstein guidelines and a common secondary or primary outcome in clinical resuscitation studies.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Rea, MD, Principal Investigator — University of Washington
Locations (1):
- King County EMS, Seattle, Washington, United States